CLINICAL TRIAL: NCT03770819
Title: Photodynamic Therapy Using Zinc Oxide Photosensitizer As An Adjunct To Scaling And Root Planing In The Management Of Chronic Periodontitis - A Split Mouth Double Blind Randomized Controlled Clinical Trial.
Brief Title: PDT As An Adjunct To SRP In The Management of Chronic Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: KLE Society's Institute of Dental Sciences (Other)
Collaborators: University of Mysore (Other)
Responsible Party: Principal Investigator, Veena H.R, Reader, Department of Periodontics, KLE Society's Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KIDSperio-PDT
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Photochemotherapy

STUDY DESIGN:
Intervention Model Description: 16 patients contributing a total of 64 sites will be selected. Recording of clinical and microbiological parameters will be done at baseline, end of 1 month, and 3 months. Oral hygiene instructions will be given. Following full mouth SRP, each quadrant will be randomly assigned by simple randomization using a computer generated randomization technique into one of the following four treatment modalities.
  Group 1 (control) - Application of placebo gel followed by sham PDT (Directing the Light cure device without turning on the light beam).
  Group 2 -Application of Zinc oxide gel followed by sham PDT. Group 3 - Application of placebo gel followed by PDT. Group 4 - Application of Zinc oxide gel followed by PDT. The procedure mentioned for each group will be performed on all periodontal pockets in the assigned quadrant at baseline, end of 1 week and 1 month from the first session.
  Study period - 3 months
Who Masked: Participant, Care Provider
Masking Description: This is a Split Mouth Double Blind Randomized Controlled Clinical Trial in which both participants and care provider are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo group (Placebo Comparator): Application of placebo gel followed by sham Photodynamic therapy
  Interventions: Procedure: Photodynamic therapy
- Zinc oxide gel group (Active Comparator): Application of Zinc oxide gel followed by sham Photodynamic therapy.
  Interventions: Procedure: Photodynamic therapy
- PDT group (Experimental): Application of placebo gel followed by Photodynamic therapy.
  Interventions: Procedure: Photodynamic therapy
- Zinc oxide and PDT group (Experimental): Application of Zinc oxide gel followed by Photodynamic therapy.
  Interventions: Procedure: Photodynamic therapy

INTERVENTIONS:
Procedure: Photodynamic therapy — Zinc oxide gel/placebo gel will be placed into the periodontal pockets using a blunt cannula ensuring that starting from the bottom, it completely fills the periodontal pockets. The gel will be retained in the pocket for 5 minutes. The perio tip will be attached to the hand piece of the light cure unit (Wavelength: 420-480nm. Light power: 1200mw/cm2 in continuous mode) and light will be activated for 60 seconds. Following this, the pockets will be irrigated with normal saline solution (0.9%Sodium chloride).
  For groups 1 and 2, sham PDT will be performed by directing the Light cure device without turning on the light beam.

SUMMARY:
The present study aims to evaluate photodynamic therapy (PDT) using Zinc oxide as a photosensitizer as an adjunct to scaling and root planing (SRP) in the management of chronic periodontitis.

DETAILED DESCRIPTION:
Following full mouth SRP, each quadrant will be randomly assigned by simple randomization using a computer generated randomization technique into one of the following four treatment modalities.

Group 1 (control) - Application of placebo gel followed by sham PDT (Directing the Light cure device without turning on the light beam).

Group 2 -Application of Zinc oxide gel followed by sham PDT. Group 3 - Application of placebo gel followed by PDT. Group 4 - Application of Zinc oxide gel followed by PDT. The procedure mentioned for each group will be performed on all periodontal pockets in the assigned quadrant at baseline, end of 1 week and 1 month from the first session.

Clinical parameters and microbial profile will be recorded at baseline (before commencement of Periodontal treatment), end of 1 month and end of 3 months following periodontal treatment.

Zinc oxide gel/placebo gel will be placed into the periodontal pockets using a blunt cannula ensuring that starting from the bottom, it completely fills the periodontal pockets. The gel will be retained in the pocket for 5 minutes. The perio tip will be attached to the hand piece of the light cure unit (Wavelength: 420-480nm. Light power: 1200mw/cm2 in continuous mode) and light will be activated for 60 seconds. Following this, the pockets will be irrigated with normal saline solution (0.9%Sodium chloride).

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders diagnosed with chronic periodontitis in the age group of 30 to 50 years with good systemic health.
* Presence of a minimum of 20 teeth and at least one site with probing pocket depth (PPD) of 4-7 mm and clinical attachment level (CAL) of 2 mm or greater, in each of the four quadrants.

Exclusion Criteria:

* Patients who have undergone periodontal therapy during the previous 6 months of commencement of the study.
* Subjects on antibiotics or immunosuppressant medication 6 months prior to the study.
* Chronic Smokers, Alcoholics, Smokeless tobacco users.
* Subjects with acute illnesses/acute intraoral lesions.
* Pregnant women and lactating mothers.
* Medically compromised subjects.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Change in Microbial profile | 3 months
  Change in levels of P.gingivalis following PDT

SECONDARY OUTCOMES:
Change in Plaque index score | 3 months
  Change in plaque index score from Range: 2-3 to Range: 0 to1.9 following PDT
Change in Gingival index score | 3 months
  Change in Gingival index score from Range: 2-3 to Range: 0 to1.9 following PDT
Probing pocket depth | 3 months
  Change in probing pocket depth from 5-7 mm to 2.9- 4.2 mm following PDT
Clinical attachment level | 3 months
  Gain in clinical attachment level following PDT

IPD SHARING:
Plan to Share IPD: Undecided